CLINICAL TRIAL: NCT01384656
Title: Effect of Glucose-insulin-potassium Solution on Myocardial Protection During Off-pump Coronary Bypass Surgery in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2009-0689
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — glucose-insulin-potassium cardioplegic solution; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GIK group (Experimental)
  Interventions: Drug: GIK solution
- Control group (Placebo Comparator)
  Interventions: Drug: GIK solution

INTERVENTIONS:
Drug: GIK solution — Patients receive 0.3 ml/kg/hr GIK solution or the same volume of normal saline depending on the group during off-pump coronary bypass surgery. GIK solution consist of 50% glucose, potassium 80 mEq, and regular insulin 325 IU/500ml.
  Other Names: glucose-insulin-potassium(GIK) solution

SUMMARY:
Patients undergoing multivessel off-pump coronary bypass surgery (OPCAB) inevitably experience cumulative ischemia-reperfusion injury at myocardium. Glucose-insulin-potassium (GIK) is a potentially useful adjunct to myocardial protection. This study was designed to evaluate the effects of GIK infusion on myocardium in patients undergoing OPCAB. Patients undergoing OPCAB with acute coronary syndrome are randomly assigned to GIK or Control group. The trial is double-blind and conducted at a single center.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing isolated OPCAB.
* Age: 20~75.

Exclusion Criteria:

* Emergency operation.
* Patients with MR ≥ 2.
* Patients with IDDM.
* Patients with random sugar ≥ 250 mg/dL.
* Patients with serum creatinine ≥ 2.0 mg/dL.
* Patients with acute myocardial infarction within 1 week of surgery

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
CK-MB(creatinine kinase-MB) mass | 12 hours after the surgery
  Comparison of cardiac enzyme elevation after surgery between GIK and Control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shim JK, Yang SY, Yoo YC, Yoo KJ, Kwak YL. Myocardial protection by glucose-insulin-potassium in acute coronary syndrome patients undergoing urgent multivessel off-pump coronary artery bypass surgery. Br J Anaesth. 2013 Jan;110(1):47-53. doi: 10.1093/bja/aes324. Epub 2012 Sep 17. PMID 22986417